CLINICAL TRIAL: NCT00426803
Title: Randomised, Double-Blind, Placebo-Controlled, Multi-centre, Parallel Groups, Study to Evaluate the Efficacy and Safety of Activated Recombinant Factor VII (NovoSeven®) in Acute Intracerebral Haemorrhage
Brief Title: Recombinant Factor VIIa in Acute Intracerebral Haemorrhage
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: F7ICH-1371
Record Dates: First submitted 2007-01-24; First posted 2007-01-25 (Estimated); Last update posted 2017-01-18 (Estimated); Status verified 2017-01

CONDITIONS: Acquired Bleeding Disorder; Intracerebral Haemorrhage
MeSH Terms: conditions — Cerebral Hemorrhage

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: activated recombinant human factor VII

SUMMARY:
This trial is conducted in North America, Europe, Asia and Oceania. The purpose of this study is to evaluate safety and efficacy of Recombinant Factor VIIa in patients with acute intracerebral bleeding.

ELIGIBILITY:
Inclusion Criteria:

* Spontaneous intracranial haemorrhage (ICH) within 3 hours after first symptom

Exclusion Criteria:

* Patients with secondary ICH
* Pre-existing disability
* Haemophilia

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Actual)
Dates: Start 2002-08; Primary Completion 2004-06 (Actual); Study Completion 2004-06 (Actual)

PRIMARY OUTCOMES:
Reducing haematoma growth

SECONDARY OUTCOMES:
Reducing disability and improving clinical outcome

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (15):
- Novo Nordisk Investigational Site, Melbourne, Australia
- Novo Nordisk Investigational Site, Graz, Austria
- Novo Nordisk Investigational Site, Antwerp, Belgium
- Novo Nordisk Investigational Site, Calgary, Canada
- Novo Nordisk Investigational Site, Aarhus, Denmark
- Novo Nordisk Investigational Site, Helsinki, Finland
- Novo Nordisk Investigational Site, Leipzig, Germany
- Novo Nordisk Investigational Site, Perugia, Italy
- Novo Nordisk Investigational Site, Amsterdam, Netherlands
- Novo Nordisk Investigational Site, Bergen, Norway
- Novo Nordisk Investigational Site, Singapore, Singapore
- Novo Nordisk Investigational Site, Madrid, Spain
- Novo Nordisk Investigational Site, Stockholm, Sweden
- Novo Nordisk Investigational Site, Lausanne, Switzerland
- Novo Nordisk Investigational Site, Newcastle upon Tyne, United Kingdom

REFERENCES:
- [Result] Mayer SA, Brun NC, Begtrup K, Broderick J, Davis S, Diringer MN, Skolnick BE, Steiner T; Recombinant Activated Factor VII Intracerebral Hemorrhage Trial Investigators. Recombinant activated factor VII for acute intracerebral hemorrhage. N Engl J Med. 2005 Feb 24;352(8):777-85. doi: 10.1056/NEJMoa042991. PMID 15728810
- [Result] Davis SM, Broderick J, Hennerici M, Brun NC, Diringer MN, Mayer SA, Begtrup K, Steiner T; Recombinant Activated Factor VII Intracerebral Hemorrhage Trial Investigators. Hematoma growth is a determinant of mortality and poor outcome after intracerebral hemorrhage. Neurology. 2006 Apr 25;66(8):1175-81. doi: 10.1212/01.wnl.0000208408.98482.99. PMID 16636233
- [Result] Steiner T, Diringer MN, Schneider D, Mayer SA, Begtrup K, Broderick J, Skolnick BE, Davis SM. Dynamics of intraventricular hemorrhage in patients with spontaneous intracerebral hemorrhage: risk factors, clinical impact, and effect of hemostatic therapy with recombinant activated factor VII. Neurosurgery. 2006 Oct;59(4):767-73; discussion 773-4. doi: 10.1227/01.NEU.0000232837.34992.32. PMID 17038942
- [Result] Zimmerman RD, Maldjian JA, Brun NC, Horvath B, Skolnick BE. Radiologic estimation of hematoma volume in intracerebral hemorrhage trial by CT scan. AJNR Am J Neuroradiol. 2006 Mar;27(3):666-70. PMID 16552014
- [Result] Broderick JP, Diringer MN, Hill MD, Brun NC, Mayer SA, Steiner T, Skolnick BE, Davis SM; Recombinant Activated Factor VII Intracerebral Hemorrhage Trial Investigators. Determinants of intracerebral hemorrhage growth: an exploratory analysis. Stroke. 2007 Mar;38(3):1072-5. doi: 10.1161/01.STR.0000258078.35316.30. Epub 2007 Feb 8. PMID 17290026
- [Result] Diringer MN, Ferran JM, Broderick J, Davis S, Mayer SA, Steiner T, Brun NC, Skolnick BE, Christensen MC. Impact of recombinant activated factor VII on health-related quality of life after intracerebral hemorrhage. Cerebrovasc Dis. 2007;24(2-3):219-25. doi: 10.1159/000104481. Epub 2007 Jun 28. PMID 17630481
- [Result] Hsia CC, Chin-Yee IH, McAlister VC. Use of recombinant activated factor VII in patients without hemophilia: a meta-analysis of randomized control trials. Ann Surg. 2008 Jul;248(1):61-8. doi: 10.1097/SLA.0b013e318176c4ec. PMID 18580208
- [Derived] Eilertsen H, Menon CS, Law ZK, Chen C, Bath PM, Steiner T, Desborough MJ, Sandset EC, Sprigg N, Al-Shahi Salman R. Haemostatic therapies for stroke due to acute, spontaneous intracerebral haemorrhage. Cochrane Database Syst Rev. 2023 Oct 23;10(10):CD005951. doi: 10.1002/14651858.CD005951.pub5. PMID 37870112
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com